CLINICAL TRIAL: NCT03213210
Title: Clinical Efficacy of Easy-graft CLASSIC for the Treatment of Peri-implantitis
Brief Title: Efficacy of Synthetic Bone Graft for Treatment of Peri-implantitis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient recruitment
Sponsor: Sunstar Americas (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLP-2017-02-18-1
Record Dates: First submitted 2017-07-07; First posted 2017-07-11 (Actual); Results first posted 2021-02-23 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-03

CONDITIONS: Peri-Implantitis
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Device treatment (Other): easy-graft CLASSIC (beta-Tricalcium Phosphate) grafting covered with polylactide membrane
  Interventions: Device: easy-graft CLASSIC (beta-Tricalcium Phosphate)

INTERVENTIONS:
Device: easy-graft CLASSIC (beta-Tricalcium Phosphate) — easy-graft will be grafted to the bone defect supporting a dental implant and covered by polylactide membrane to facilitate regeneration of new bone and healthy attachment to stabilize the dental implant.
  Other Names: GUIDOR Bioresorbable Matrix Barrier

SUMMARY:
Single arm study to evaluate the effectiveness of treatment approach using a new moldable beta-tricalcium phosphate(TCP) bone graft material and polylactide membrane in peri-implantitis.

ELIGIBILITY:
Inclusion Criteria:

* Subject has read and signed the Institutional Review Board approved consent form before treatment.
* Subject must be age 21 or above.
* Subject must be willing and able to follow study procedures and instructions.
* Subject affected by moderate to severe peri-implant disease.
* Treated chronic periodontitis and proper periodontal maintenance care.
* Dental implant must meet the following criteria to be selected for the study:

  1. Implant presenting Probing Depth ≥ 6 mm
  2. Radiographic implant bone loss more than 25% of the implant length (Apex of the implant to implant platform) .
  3. Peri implant bone defect being a buccal dehiscence and semicircular bone resorption to the middle of the implant body, buccal dehiscence and circular bone resorption with lingual bone plate intact or circular bone resorption with buccal and lingual bone plates intact
  4. Single tooth implant restoration or implant supported fixed partial denture.

Exclusion Criteria:

* Subjects participating (currently or within 30 days prior to enrollment) in other clinical trials involving therapeutic intervention (either medical or dental).
* Subjects with poor oral hygiene as indicated by a score of greater than 50% on the O'Leary Plaque Index.
* Subjects with a systemic condition, which would preclude periodontal treatment, including but not limited to uncontrolled diabetes.
* Subjects with acute infectious lesions in the areas intended for treatment.
* Subjects taking chronic (i.e., > 2 weeks), therapeutic doses of medications known to affect bone metabolism such as nonsteroidal anti-inflammatory drugs or bisphosphonates. Prophylactic aspirin (≤ 325 mg q.d.) for cardiovascular indications will be permitted in subjects.
* Female subjects who are pregnant or lactating, or sexually-active female subjects who are of childbearing potential and are not using hormonal or barrier methods of birth control. (except for when a result of pregnancy test is negative)
* Subjects who are on any chronic antibiotic or steroidal therapy.
* Smoker using more than 10 cigarettes or equivalent per day.
* Smoker using cigar, smokeless tobacco use or e-cigarette.
* Subjects diagnosed with drug induced gingival hyperplasia (e.g. calcium channel blockers).
* Subjects with radiographic evidence of pathology in other areas of the mouth besides implant area to be treated.
* Implant mobility.
* Subjects with parafunctional habits and not wearing bite guard.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-11-12 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-01-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Creighton University School of Dentisty, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Device Treatment
Started | 5
6-month Follow-up | 3
Completed | 0
Not Completed | 5
Not completed — Lost to Follow-up | 2
Not completed — Study termination | 3

BASELINE CHARACTERISTICS:
Arm/Group | Device Treatment
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.6 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Probing Depth
Description: Distance of probe penetration from gingival margin to bottom of peri-implant pocket
Time Frame: Change from baseline at 12 months after the surgery
Population: No subjects were examined at 12 months after the surgery.
Arm/Group | Device Treatment
Number analyzed (Participants) | 0

2. Primary Outcome: Esthetic Satisfaction
Description: To be assessed by examiner and subject using the Visual Analog Scales
Time Frame: At 12 months after the surgery
Population: No subjects were examined at 12 months after the surgery.
Arm/Group | Device Treatment
Number analyzed (Participants) | 0

3. Secondary Outcome: Change of Marginal Bone Level
Description: Change of marginal bone level on periapical standardized radiographs from baseline.
Time Frame: Change from baseline at 6 and 12 months after the surgery
Population: Marginal bone level was examined in 3 subjects at 6-month follow-up. No subjects were examined at 12 months after the surgery.
Measure: Mean (Standard Deviation); unit: percentage of bone height change
Arm/Group | Device Treatment
Number analyzed (Participants) | 3
percentage of bone height change
  6 months | 3.3 (5.8)
  12 months: number analyzed (Participants) | 0

4. Secondary Outcome: Change in Width of Keratinized Tissue
Description: Distance between free gingival margin and mucogingival junction
Time Frame: Change from baseline at 6 and 12 months after the surgery
Population: No subjects were examined at 6 and 12 months after the surgery.
Arm/Group | Device Treatment
Number analyzed (Participants) | 0

5. Secondary Outcome: Change in Clinical Attachment Level
Description: Distance of probe penetration from fixed reference to bottom of peri-implant
Time Frame: Change from baseline to at 6 and 12 months after the surgery
Population: No subjects were examined at 6 and 12 months after the surgery.
Arm/Group | Device Treatment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 6 months after the surgery
Arm/Group | Device Treatment
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-22): https://cdn.clinicaltrials.gov/large-docs/10/NCT03213210/Prot_SAP_000.pdf